CLINICAL TRIAL: NCT03598777
Title: A Phase II, Multicentre, Double-blind, Randomised, Placebo Controlled, Dose Escalation and Dose Finding Study to Evaluate the Efficacy and Safety of Dysport in Vulvodynia Patients
Brief Title: Dysport in Vulvodynia Phase II Study
Acronym: DYVINIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D-FR-52120-236
Record Dates: First submitted 2018-06-08; First posted 2018-07-26 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-10

CONDITIONS: Vulvodynia
MeSH Terms: conditions — Vulvodynia | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dysport - Dose Escalation stage 1 (Experimental): Intramuscular injection of Dysport on day 1 of each cycle.
  Interventions: Biological: Botulinum toxin type A
- Placebo - Dose Escalation stage 1 and Dose Expansion stage 2 (Placebo Comparator): Intramuscular injection on day 1 of cycle 1.
  Interventions: Drug: Placebo
- Dysport - Dose Expansion stage 2 (Active Comparator): Depending upon the results from Stage 1 one or two doses of Dysport will be selected. Intramuscular injection of Dysport on day 1 of each cycle.
  Interventions: Biological: Botulinum toxin type A

INTERVENTIONS:
Biological: Botulinum toxin type A — Botulinum Toxin Type A (Dysport) using a vial of 500 U will be injected intramuscularly across pelvic floor muscles.
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: Dysport - Dose Escalation stage 1; Dysport - Dose Expansion stage 2
Drug: Placebo — The reconstituted solution will be injected intramuscularly across pelvic floor muscles.
  Arms: Placebo - Dose Escalation stage 1 and Dose Expansion stage 2

SUMMARY:
This study is designed to define optimal doses of Dysport and evaluate its efficacy and safety compared with placebo for the treatment of vulvodynia.

The study will consist of a dose escalation stage (Stage 1) and a dose expansion stage (Stage 2). Both Stage 1 and Stage 2 will consist of a double-blind period (with treatment cycle 1; Dysport or placebo) followed by an open label treatment period. One or two optimally safe and effective doses of Dysport selected from Stage 1 will be further investigated in the Stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* Have vulvodynia for at least 6 months and for no more than 15 years
* Have provoked pain at the vestibule on a Q tip test

Exclusion Criteria:

* Deep pain during intercourse
* Have genitourinary or gastrointestinal conditions which may interfere with the study
* Previous surgery that according to investigator's judgement may impact on study outcome (including but not limited to hysterectomy, vestibulectomy, urologic surgery, perianal surgery) or genital trauma or mutilation/cutting

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (9):
- United States (8):
  - James A. Simon, MD, PC, Washington D.C., District of Columbia
  - The Center for Vulvovaginal Disorders, Washington D.C., District of Columbia
  - New Age Medical Research Corporation, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Missouri
  - Omaha OB-GYN Associates, PC, Omaha, Nebraska
  - The Center for Vulvovaginal Disorders, New York, New York
  - Women's Institute for Sexual Health (WISH), Nashville, Tennessee
  - Seattle Women's: Health, Research, Gynecology®, Seattle, Washington
- Clinique de Santé des Femmes, Québec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Goldstein A, Rubin R, Dahir M, Goldstein I, Faught BM, Bohm-Starke N, Krapf J, Caetano P, Volteau M, Silva R. Phase 2 randomized study of abobotulinumtoxinA in patients with provoked vestibulodynia: dose-finding results. J Sex Med. 2025 Apr 15;22(4):588-596. doi: 10.1093/jsxmed/qdaf022. PMID 39953376

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase II double-blind (DB) study was conducted in participants with vulvodynia provoked vestibulodynia. 8 sites in the United States and Canada randomised participants. The study consisted of a dose escalation stage (Stage 1) and a dose expansion stage (Stage 2). The purpose of the dose escalation (Stage 1) was to determine the Dysport doses to be further investigated in Stage 2. All analysis was based on available Stage 1 data only. Stage 2 was not started due to early study termination.
Pre-assignment Details: For each participant, the study consisted of a DB treatment period (Cycle 1; participants received Dysport or placebo) followed by a follow-up period and/or open-label (OL) treatment period (Cycles 2 to 4; participants received Dysport). A total of 60 participants were randomised and received treatment with placebo or Dysport in the DB treatment period for Stage 1. Up to a maximum of 800 Units (U) Dysport was planned but 500 U was the maximum dose tested due to early study termination.
Groups:
- Placebo: Stage 1: On Cycle 1 Day 1 in the DB treatment period, participants received placebo (matching with Dysport) injected intramuscularly at 10 injection sites across 4 pelvic floor muscles in the vestibular region.
  Following Week 12 of the DB treatment period, all participants who met retreatment criteria were treated during the OL period for Cycles 2 to 4 (with each treatment administered at least 12 weeks apart). For a given participant, the Dysport dose during the OL treatment period was based on the investigator's judgement (based on efficacy and safety).
- Dysport 100 U: Stage 1: On Cycle 1 Day 1 in the DB treatment period, participants received Dysport 100 U injected intramuscularly at 10 injection sites across 4 pelvic floor muscles in the vestibular region.
  Following Week 12 of the DB treatment period, all participants who met retreatment criteria were treated during the OL period for Cycles 2 to 4 (with each treatment administered at least 12 weeks apart). For a given participant, the Dysport dose during the OL treatment period was based on the investigator's judgement (based on efficacy and safety).
- Dysport 300 U: Stage 1: On Cycle 1 Day 1 in the DB treatment period, participants received Dysport 300 U injected intramuscularly at 10 injection sites across 4 pelvic floor muscles in the vestibular region.
  Following Week 12 of the DB treatment period, all participants who met retreatment criteria were treated during the OL period for Cycles 2 to 4 (with each treatment administered at least 12 weeks apart). For a given participant, the Dysport dose during the OL treatment period was based on the investigator's judgement (based on efficacy and safety).
- Dysport 400 U: Stage 1: On Cycle 1 Day 1 in the DB treatment period, participants received Dysport 400 U injected intramuscularly at 10 injection sites across 4 pelvic floor muscles in the vestibular region.
  Following Week 12 of the DB treatment period, all participants who met retreatment criteria were treated during the OL period for Cycles 2 to 4 (with each treatment administered at least 12 weeks apart). For a given participant, the Dysport dose during the OL treatment period was based on the investigator's judgement (based on efficacy and safety).
- Dysport 500 U: Stage 1: On Cycle 1 Day 1 in the DB treatment period, participants received Dysport 500 U injected intramuscularly at 10 injection sites across 4 pelvic floor muscles in the vestibular region.
  Following Week 12 of the DB treatment period, all participants who met retreatment criteria were treated during the OL period for Cycles 2 to 4 (with each treatment administered at least 12 weeks apart). For a given participant, the Dysport dose during the OL treatment period was based on the investigator's judgement (based on efficacy and safety).
Period: Overall Study
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
Started | 13 | 8 | 8 | 14 | 17
Received Treatment in Cycle 1 DB Treatment Period | 13 | 8 | 8 | 14 | 17
Retreated in Cycle 2 OL Treatment Period | 13 | 7 | 8 | 13 | 11
Retreated in Cycle 3 OL Treatment Period | 8 | 6 | 6 | 12 | 2
Retreated in Cycle 4 OL Treatment Period | 1 | 0 | 1 | 3 | 0
Completed | 7 | 7 | 8 | 14 | 2
Not Completed | 6 | 1 | 0 | 0 | 15
Not completed — Study Terminated by Sponsor | 3 | 0 | 0 | 0 | 15
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomised participants were included in the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U | Total
Number analyzed (Participants) | 13 | 8 | 8 | 14 | 17 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 8 | 8 | 14 | 17 | 60
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (7.12) | 29.6 (3.11) | 30.4 (6.61) | 31.1 (5.00) | 26.5 (5.48) | 29.4 (5.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 8 | 14 | 17 | 60
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants may have more than one race.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
    Asian | 1 | 0 | 0 | 0 | 1 | 2
    Black or African American | 0 | 0 | 0 | 1 | 1 | 2
    White | 12 | 7 | 8 | 13 | 15 | 55
    Other | 0 | 2 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 1 | 4
  Not Hispanic or Latino | 11 | 8 | 8 | 13 | 16 | 56
Dilator Maximum Tested Size (DMTS) at Baseline [Mean (Standard Deviation); unit: scores on a scale] — A set of 8 vaginal dilators of increasing diameter (#1 being the smallest and #8 being the largest) were used by the investigator to provoke pain to allow assessment of vestibular pain intensity in each participant. Participants rated the pain for each dilator size on an 11-point Numeric Rating Scale (NRS) ranging from 0 to 10, where 0 was no pain and 10 was the worst possible pain. Higher scores indicate a worse outcome. Based on the subjective pain threshold, the largest sized dilator that the participant accepted/tolerated for the test was defined as the DMTS at the Baseline visit.
  scores on a scale | 4.5 (1.27) | 4.4 (1.19) | 4.8 (1.04) | 4.5 (1.02) | 4.1 (1.11) | 4.4 (1.11)
Pain reported using DMTS at Baseline [Mean (Standard Deviation); unit: scores on a scale] — A set of 8 vaginal dilators of increasing diameter (#1 being the smallest and #8 being the largest) were used by the investigator to provoke pain to allow assessment of vestibular pain intensity in each participant. Participants rated the pain for each dilator size on an 11-point NRS ranging from 0 to 10, where 0 was no pain and 10 was the worst possible pain. Higher scores indicate a worse outcome. Based on the subjective pain threshold, the largest sized dilator that the participant accepted/tolerated for the test was defined as the DMTS at the Baseline visit.
  scores on a scale | 7.2 (1.83) | 6.5 (0.93) | 7.4 (1.60) | 6.3 (0.99) | 7.4 (1.00) | 7.0 (1.34)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) During the DB Treatment Period (Stage 1)
Description: For Stage 1, the primary endpoint was safety during the DB treatment period as assessed by the incidence of adverse events (AEs). An AE was the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition could have been symptoms, signs or abnormal results of an investigation. A TEAE was an event with start date on or after the date of the first investigational medicinal product (IMP). Relatedness to treatment was assessed by the investigator. TEAEs of special interest included events suggesting a possible remote spread of effect of the toxin, events related to urinary incontinence or faecal incontinence and events assessed as a potential hypersensitivity reaction. Results for this outcome are reported as the number of participants experiencing at least one TEAE in each specified category.
Time Frame: From Baseline (Cycle 1 Day 1) to Cycle 1 Week 12 (DB treatment period, Stage 1)
Population: The safety population included all randomised participants who received at least one IMP administration (including only partial administration).
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Stage 1: On Cycle 1 Day 1 in the DB treatment period, participants received placebo (matching with Dysport) injected intramuscularly at 10 injection sites across 4 pelvic floor muscles in the vestibular region.
- Dysport 100 U: Stage 1: On Cycle 1 Day 1 in the DB treatment period, participants received Dysport 100 U injected intramuscularly at 10 injection sites across 4 pelvic floor muscles in the vestibular region.
- Dysport 300 U: Stage 1: On Cycle 1 Day 1 in the DB treatment period, participants received Dysport 300 U injected intramuscularly at 10 injection sites across 4 pelvic floor muscles in the vestibular region.
- Dysport 400 U: Stage 1: On Cycle 1 Day 1 in the DB treatment period, participants received Dysport 400 U injected intramuscularly at 10 injection sites across 4 pelvic floor muscles in the vestibular region.
- Dysport 500 U: Stage 1: On Cycle 1 Day 1 in the DB treatment period, participants received Dysport 500 U injected intramuscularly at 10 injection sites across 4 pelvic floor muscles in the vestibular region.
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
Number analyzed (Participants) | 13 | 8 | 8 | 14 | 17
Participants
  Any TEAEs | 1 | 3 | 3 | 3 | 6
  Severe TEAEs | 0 | 0 | 0 | 0 | 0
  Treatment-related TEAEs | 1 | 0 | 0 | 0 | 3
  TEAEs leading to IMP withdrawal | 0 | 0 | 0 | 0 | 0
  Serious AEs | 0 | 0 | 0 | 0 | 0
  TEAEs leading to death | 0 | 0 | 0 | 0 | 0
  TEAEs of special interest | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Mean Change From Baseline in Vaginal Dilator Induced Pain During the DB Treatment Period at Week 6 (Stage 2)
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 1 Week 6 (DB treatment period, Stage 2)
Population: The study was terminated early prior to starting Stage 2; therefore no analysis was performed for this primary outcome.
Groups:
- Placebo: Stage 2: On Cycle 1 Day 1 in the DB treatment period, participants were to receive placebo (matching with Dysport) injected intramuscularly at 10 injection sites across 4 pelvic floor muscles in the vestibular region.
- Dysport High Dose: Stage 2: On Cycle 1 Day 1 in the DB treatment period, participants were to receive Dysport high dose, corresponding to the optimal highest safe and efficacious dose selected from Stage 1, injected intramuscularly at 10 injection sites across 4 pelvic floor muscles in the vestibular region.
- Dysport Low Dose: Stage 2: On Cycle 1 Day 1 in the DB treatment period, participants were to receive Dysport low dose, selected based on safety and efficacy considerations observed in Stage 1, injected intramuscularly at 10 injection sites across 4 pelvic floor muscles in the vestibular region.
Arm/Group | Placebo | Dysport High Dose | Dysport Low Dose
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Mean Change From Baseline in Vaginal Dilator Induced Pain as Reported on an 11-point Numeric Rating Scale (NRS) During the DB Treatment Period at Week 6 and Week 12 (Stage 1)
Description: For the dilator test, a vaginal dilator was used by the investigator to provoke pain to allow assessment of vestibular pain intensity in each participant. Participants rated their pain using an 11-point NRS ranging from 0 to 10, where 0 was no pain and 10 was the worst possible pain. Higher scores indicate a worse outcome. The dilator test was used to assess the change from Baseline in the vaginal dilator induced pain (using the DMTS reported at Baseline). Baseline was defined as the last value available prior to the first study IMP treatment administration. Results for this outcome are reported as change from Baseline during the DB treatment period at Week 6 and Week 12.
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 1 Week 6 and Week 12 (DB treatment period, Stage 1)
Population: The modified Intent-To-Treat population (mITT) included all randomised participants who received at least one IMP administration and had data for the vaginal dilator induced pain as reported on an 11-point NRS at Baseline and Cycle 1 Week 6 visit. Only participants with values at both Baseline and the specified visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
Number analyzed (Participants) | 13 | 8 | 8 | 14 | 17
scores on a scale
  Week 6 | -3.3 (3.01) | -2.4 (2.26) | -4.1 (3.68) | -1.9 (2.62) | -2.1 (2.56)
  Week 12 | -3.2 (2.76) | -2.8 (3.01) | -4.1 (3.44) | -1.8 (2.29) | -2.7 (2.08)

4. Secondary Outcome: Number of Participants Who Reported at Least a 50% Decrease From Baseline in Vaginal Dilator Induced Pain as Reported on an 11-point NRS During the DB Treatment Period at Week 6 and Week 12 (Stage 1)
Description: For the dilator test, a vaginal dilator was used by the investigator to provoke pain to allow assessment of vestibular pain intensity in each participant. Participants rated their pain using an 11-point NRS ranging from 0 to 10, where 0 was no pain and 10 was the worst possible pain. Higher scores indicate a worse outcome. The dilator test was used to assess the change from Baseline in the vaginal dilator induced pain (using the DMTS reported at Baseline). Baseline was defined as the last value available prior to the first study IMP treatment administration. Results for this outcome are reported as the number of participants who had a ≥50% decrease from Baseline during the DB treatment period at Week 6 and Week 12.
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 1 Week 6 and Week 12 (DB treatment period, Stage 1)
Population: The mITT population included all randomised participants who received at least one IMP administration and had data for the vaginal dilator induced pain as reported on an 11-point NRS at Baseline and Cycle 1 Week 6 visit. Only participants with values at both Baseline and the specified visit were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
Number analyzed (Participants) | 13 | 8 | 8 | 14 | 17
Participants
  Week 6 | 6 | 3 | 5 | 4 | 5
  Week 12 | 6 | 3 | 4 | 3 | 6

5. Secondary Outcome: Number of Participants Who Reported at Least a 30% Decrease From Baseline in Vaginal Dilator Induced Pain as Reported on an 11-point NRS During the DB Treatment Period at Week 6 and Week 12 (Stage 1)
Description: For the dilator test, a vaginal dilator was used by the investigator to provoke pain to allow assessment of vestibular pain intensity in each participant. Participants rated their pain using an 11-point NRS ranging from 0 to 10, where 0 was no pain and 10 was the worst possible pain. Higher scores indicate a worse outcome. The dilator test was used to assess the change from Baseline in the vaginal dilator induced pain (using the DMTS reported at Baseline). Baseline was defined as the last value available prior to the first study IMP treatment administration. Results for this outcome are reported as the number of participants who had a ≥30% decrease from Baseline during the DB treatment period at Week 6 and Week 12.
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 1 Week 6 and Week 12 (DB treatment period, Stage 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
Number analyzed (Participants) | 13 | 8 | 8 | 14 | 17
Participants
  Week 6 | 9 | 4 | 5 | 10 | 7
  Week 12 | 7 | 3 | 5 | 8 | 10

6. Secondary Outcome: Number of Participants Who Reported at Least a 2-point Decrease From Baseline in Vaginal Dilator Induced Pain as Reported on an 11-point NRS During the DB Treatment Period at Week 6 and Week 12 (Stage 1)
Description: For the dilator test, a vaginal dilator was used by the investigator to provoke pain to allow assessment of vestibular pain intensity in each participant. Participants rated their pain using an 11-point NRS ranging from 0 to 10, where 0 was no pain and 10 was the worst possible pain. Higher scores indicate a worse outcome. The dilator test was used to assess the change from Baseline in the vaginal dilator induced pain (using the DMTS reported at Baseline). Baseline was defined as the last value available prior to the first study IMP treatment administration. Results for this outcome are reported as the number of participants who had a ≥2-point decrease from Baseline during the DB treatment period at Week 6 and Week 12.
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 1 Week 6 and Week 12 (DB treatment period, Stage 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
Number analyzed (Participants) | 13 | 8 | 8 | 14 | 17
Participants
  Week 6 | 9 | 5 | 6 | 10 | 9
  Week 12 | 10 | 5 | 6 | 8 | 12

7. Secondary Outcome: Mean Change From Baseline in the DTMS During the DB Treatment Period at Week 6 and Week 12 (Stage 1)
Description: For the dilator test, a set of 8 vaginal dilators of increasing diameter (#1 being the smallest and #8 being the largest) were used by the investigator to provoke pain to allow assessment of vestibular pain intensity in each participant. Based on the subjective pain threshold, the largest sized dilator that the participant accepted/tolerated for the test, was defined as the DMTS. Participants rated their pain using an 11-point NRS ranging from 0 to 10, where 0 was no pain and 10 was the worst possible pain. Higher scores indicate a worse outcome. Baseline was defined as the last value available prior to the first study IMP treatment administration. Results for this outcome are reported as change from Baseline in the DTMS during the DB treatment period at Week 6 and Week 12.
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 1 Week 6 and Week 12 (DB treatment period, Stage 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
Number analyzed (Participants) | 13 | 8 | 8 | 14 | 17
scores on a scale
  Week 6 | 1.5 (1.27) | 1.3 (1.04) | 1.6 (1.19) | 1.4 (1.45) | 1.4 (1.46)
  Week 12 | 1.0 (1.00) | 1.4 (1.06) | 1.8 (1.49) | 1.1 (1.64) | 1.5 (1.42)

8. Secondary Outcome: Mean Change From Baseline in the Composite Score for the Vaginal Dilator Induced Pain and Dilator Size During the DB Treatment Period at Week 6 and Week 12 (Stage 1)
Description: For the dilator test, a set of 8 vaginal dilators of increasing diameter (#1 being the smallest and #8 being the largest) were used by the investigator to provoke pain to allow assessment of vestibular pain intensity in each participant. The composite score for the vaginal dilator induced pain and dilator size was the sum of all pain measurements across the full range of dilator sizes. For any dilator size that was beyond the DMTS, the pain score was 10. There was to be at least 6 pain scores (recorded by the investigator) to calculate the composite score. Participants rated their pain using an 11-point NRS ranging from 0 to 10, where 0 was no pain and 10 was the worst possible pain. Higher scores indicate a worse outcome. Baseline was defined as the last value available prior to the first study IMP treatment administration. Results for this outcome are reported as change from Baseline in the composite score for the dilator test during the DB treatment period at Week 6 and Week 12.
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 1 Week 6 and Week 12 (DB treatment period, Stage 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
Number analyzed (Participants) | 13 | 8 | 8 | 14 | 17
scores on a scale
  Week 6 | -15.1 (11.16) | -13.0 (12.90) | -24.4 (15.97) | -13.4 (15.59) | -11.5 (15.09)
  Week 12 | -12.2 (10.52) | -14.0 (14.66) | -23.6 (18.09) | -11.6 (12.60) | -13.7 (15.02)

9. Secondary Outcome: Mean Change From Baseline in Pain During Insertion of Vaginal Dilator Number 6 Size as Reported on an 11-point NRS During the DB Treatment Period at Week 6 and Week 12 (Stage 1)
Description: From 2 weeks prior to the next planned visit, all participants rated in the electronic diary (eDiary) once a week the level of the corresponding pain following insertion of the number 6 vaginal dilator into the vagina. Participants rated their pain using an 11-point NRS ranging from 0 to 10, where 0 was no pain and 10 was the worst possible pain. Higher scores indicate a worse outcome. Baseline was defined as the last value available prior to the first study IMP treatment administration. Results for this outcome are reported as the change from Baseline in participant reported pain score for the number 6 dilator test during the DB treatment period at Week 6 and Week 12.
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 1 Week 6 and Week 12 (DB treatment period, Stage 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
Number analyzed (Participants) | 10 | 7 | 6 | 14 | 16
scores on a scale
  Week 6: number analyzed (Participants) | 8 | 6 | 6 | 12 | 16
  Week 6 | -2.69 (2.549) | -1.75 (2.340) | -2.17 (2.893) | -1.50 (1.871) | -1.94 (1.841)
  Week 12: number analyzed (Participants) | 10 | 6 | 5 | 12 | 13
  Week 12 | -2.10 (1.983) | -1.17 (2.503) | -2.80 (2.280) | -1.04 (1.196) | -2.38 (1.949)

10. Secondary Outcome: Number of Participants Who Reported at Least a 50% Decrease From Baseline in Pain During Insertion of Vaginal Dilator Number 6 Size as Reported on an 11-point NRS During the DB Treatment Period at Week 6 and Week 12 (Stage 1)
Description: From 2 weeks prior to the next planned visit, all participants rated in the eDiary once a week the level of the corresponding pain following insertion of the number 6 vaginal dilator into the vagina. Participants rated their pain using an 11-point NRS ranging from 0 to 10, where 0 was no pain and 10 was the worst possible pain. Higher scores indicate a worse outcome. Baseline was defined as the last value available prior to the first study IMP treatment administration. Results for this outcome are reported as the number of participants who had a ≥50% decrease from Baseline in participant reported pain score for the number 6 dilator test during the DB treatment period at Week 6 and Week 12.
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 1 Week 6 and Week 12 (DB treatment period, Stage 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
Number analyzed (Participants) | 13 | 8 | 8 | 14 | 17
Participants
  Week 6: number analyzed (Participants) | 8 | 6 | 6 | 12 | 16
  Week 6 | 3 | 1 | 2 | 2 | 4
  Week 12: number analyzed (Participants) | 10 | 6 | 5 | 12 | 13
  Week 12 | 4 | 1 | 2 | 2 | 4

11. Secondary Outcome: Number of Participants Who Reported at Least a 30% Decrease From Baseline in Pain During Insertion of Vaginal Dilator Number 6 Size as Reported on an 11-point NRS During the DB Treatment Period at Week 6 and Week 12 (Stage 1)
Description: From 2 weeks prior to the next planned visit, all participants rated in the eDiary once a week the level of the corresponding pain following insertion of the number 6 vaginal dilator into the vagina. Participants rated their pain using an 11-point NRS ranging from 0 to 10, where 0 was no pain and 10 was the worst possible pain. Higher scores indicate a worse outcome. Baseline was defined as the last value available prior to the first study IMP treatment administration. Results for this outcome are reported as the number of participants who had a ≥30% decrease from Baseline in participants reported pain score for the number 6 dilator test during the DB treatment period at Week 6 and Week 12.
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 1 Week 6 and Week 12 (DB treatment period, Stage 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
Number analyzed (Participants) | 13 | 8 | 8 | 14 | 17
Participants
  Week 6: number analyzed (Participants) | 8 | 6 | 6 | 12 | 16
  Week 6 | 5 | 3 | 2 | 3 | 8
  Week 12: number analyzed (Participants) | 10 | 6 | 5 | 12 | 13
  Week 12 | 6 | 2 | 3 | 2 | 6

12. Secondary Outcome: Number of Participants Who Reported at Least a 2-point Decrease From Baseline in Pain During Insertion of Vaginal Dilator Number 6 Size as Reported on an 11-point NRS During the DB Treatment Period at Week 6 and Week 12 (Stage 1)
Description: From 2 weeks prior to the next planned visit, all participants rated in the eDiary once a week the level of the corresponding pain following insertion of the number 6 vaginal dilator into the vagina. Participants rated their pain using an 11-point NRS ranging from 0 to 10, where 0 was no pain and 10 was the worst possible pain. Higher scores indicate a worse outcome. Baseline was defined as the last value available prior to the first study IMP treatment administration. Results for this outcome are reported as the number of participants who had a 2-point decrease from Baseline in participant reported pain score for the number 6 dilator test during the DB treatment period at Week 6 and Week 12.
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 1 Week 6 and Week 12 (DB treatment period, Stage 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
Number analyzed (Participants) | 13 | 8 | 8 | 14 | 17
Participants
  Week 6: number analyzed (Participants) | 8 | 6 | 6 | 12 | 16
  Week 6 | 5 | 3 | 2 | 3 | 8
  Week 12: number analyzed (Participants) | 10 | 6 | 5 | 12 | 13
  Week 12 | 5 | 2 | 2 | 2 | 7

13. Secondary Outcome: Mean Change From Baseline in Pain During Intercourse as Reported on an 11-point NRS During the DB Treatment Period at Week 6 and Week 12 (Stage 1)
Description: From the Screening visit, and then 2 weeks prior to the next planned visit, participants recorded on a daily basis in the eDiary if they had intercourse and if yes, the level of the corresponding pain during each intercourse instance. Participants rated their pain using an 11-point NRS ranging from 0 to 10, where 0 was no pain and 10 was the worst possible pain. Higher scores indicate a worse outcome. The 2-week average was used, which was calculated as the average of the score over the last 2 weeks (14 days) prior to the visit. Baseline was defined as the last value available prior to the first study IMP treatment administration. Results for this outcome are reported as the change from Baseline in participant reported pain score during intercourse (over the last 2 weeks prior to each visit) during the DB treatment period at Week 6 and Week 12.
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 1 Week 6 and Week 12 (DB treatment period, Stage 1)
Population: The mITT population included all randomised participants who received at least one IMP administration and had data for the vaginal dilator induced pain as reported on an 11-point NRS at Baseline and Cycle 1 Week 6 visit. Only participants who had intercourse in the corresponding period, with values at both Baseline and the specified visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 9
scores on a scale
  Week 6: number analyzed (Participants) | 2 | 3 | 6 | 6 | 8
  Week 6 | -5.68 (4.502) | -0.43 (3.092) | -2.01 (2.025) | -0.51 (2.186) | -1.91 (2.291)
  Week 12: number analyzed (Participants) | 4 | 3 | 3 | 5 | 9
  Week 12 | -3.04 (4.246) | 0.20 (2.207) | -1.58 (2.671) | -0.88 (3.206) | -2.38 (2.120)

14. Secondary Outcome: Mean Change From Baseline in the Number of Intercourse Instances in Participants With Partners During the DB Treatment Period at Week 6 and Week 12 (Stage 1)
Description: From the Screening visit, and then 2 weeks prior to the next planned visit, participants recorded on a daily basis in the eDiary if they had intercourse and if yes, the number of intercourse instances in the previous 24-hour period. The number of intercourse instances over the 2 weeks preceding the visit was calculated as the total recorded number of intercourse instances over 14 days prior to the visit. Baseline was defined as the last value available prior to the first study IMP treatment administration. Results for this outcome are reported as the change from Baseline in number of intercourse instances (over the last 2 weeks prior to each visit) during the DB treatment period at Week 6 and Week 12.
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 1 Week 6 and Week 12 (DB treatment period, Stage 1)
Population: The mITT population included all randomised participants who received at least one IMP administration and had data for the vaginal dilator induced pain as reported on an 11-point NRS at Baseline and Cycle 1 Week 6 visit. Only participants who had a partner, with values at both Baseline and the specified visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
Number analyzed (Participants) | 11 | 6 | 7 | 11 | 14
scores on a scale
  Week 6: number analyzed (Participants) | 10 | 6 | 7 | 10 | 13
  Week 6 | -1.0 (3.89) | 0.3 (3.01) | -0.1 (3.63) | -0.3 (1.25) | -1.1 (1.50)
  Week 12: number analyzed (Participants) | 10 | 5 | 6 | 11 | 12
  Week 12 | -1.3 (2.45) | -2.6 (2.88) | -1.5 (2.07) | -0.1 (1.92) | -1.5 (1.51)

15. Secondary Outcome: Use of Pain Rescue Medication Associated With Intercourse During the DB Treatment Period at Week 6 and Week 12
Description: From the Screening visit, and then 2 weeks prior to the next planned visit, participants recorded on a daily basis in the eDiary if they had intercourse and also details of any pain rescue medication consumed for each intercourse instance to prevent or treat the vestibular pain. If a participant used the rescue medication associated with at least one instance during the 2-week prior to a visit, the participant was considered as having used the rescue medication for that visit. Results for this outcome are reported as the number of participants using pain rescue medication associated with intercourse (over the last 2 weeks prior to each visit) during the DB treatment period at Baseline, Week 6 and Week 12.
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 1 Week 6 and Week 12 (DB treatment period, Stage 1)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
Number analyzed (Participants) | 7 | 5 | 7 | 9 | 10
Participants
  Baseline: number analyzed (Participants) | 6 | 4 | 6 | 6 | 9
  Baseline | 0 | 0 | 1 | 0 | 1
  Week 6: number analyzed (Participants) | 3 | 4 | 7 | 7 | 9
  Week 6 | 0 | 0 | 0 | 2 | 0
  Week 12: number analyzed (Participants) | 4 | 3 | 3 | 7 | 10
  Week 12 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs were collected from first administration of IMP (Cycle 1 Day 1) up to end of the DB treatment period; duration of 12 weeks.
Description: The safety population included all randomised participants who received at least one IMP administration (including only partial administration).
Arm/Group | Placebo | Dysport 100 U | Dysport 300 U | Dysport 400 U | Dysport 500 U
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/8 | 0/8 | 0/14 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/8 | 0/8 | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 1/13 | 3/8 | 3/8 | 3/14 | 6/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Dysport 100 U (N=8) | Dysport 300 U (N=8) | Dysport 400 U (N=14) | Dysport 500 U (N=17)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple allergies (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Retinal migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
After all participants completed Week 12, a Data Review Committee (DRC) recommended: "No safety concerns noted in review of all available data. Efficacy cannot be assessed due to the small sample size of cohorts. The DRC would recommend that Stage 1 is not used to make an efficacy assessment; therefore, there is no justification to increase the dose, nor to move to Stage 2." Thus, sponsor terminated the study early; the decision was not related to any safety/tolerability concerns with Dysport.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT03598777/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT03598777/SAP_001.pdf